CLINICAL TRIAL: NCT03532971
Title: Prospective Study of BK Virus Disease After Allogeneic Hematopoietic-cell Transplantation: Defining BK Disease's Natural History, Clinical Spectrum, Immunology, and Outcomes
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jerome Ritz, MD, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 17-664
Record Dates: First submitted 2018-05-10; First posted 2018-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: BK Virus Infection
Keywords: BK virus; BK polyomavirus; hematopoietic-cell transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- allogeneic hematopoietic-cell transplantation patients: Prospective HCT cohort of patients undergoing allogeneic HCT at DFCI
  Interventions: Other: Symptom index questionnaire; Diagnostic Test: BK polyomavirus PCR; Other: quality of life questionnaires

INTERVENTIONS:
Other: Symptom index questionnaire — A survey administered to identify the symptoms of the patient
Diagnostic Test: BK polyomavirus PCR — quantitative PCR testing
Other: quality of life questionnaires — Standard questionnaires validated for HCT recipients

SUMMARY:
This research study is evaluating the reactivation of BK virus in patients who have undergone allogeneic hematopoietic-cell transplantation.

DETAILED DESCRIPTION:
Every year, more than 25,000 patients worldwide receive lifesaving bone marrow transplantations with hematopoietic-cells from another person. It is estimated that over 75% of these patients will develop an infectious complication, of which approximately one third can be life-threatening. A significant proportion of these infections are caused by opportunistic viruses, such as BK virus.

This virus establishes latent infection in most individuals, but does not normally cause disease. It can reactivate after hematopoietic-cell transplantation and represents the second most common viral infection in this patient population. BK virus is associated with kidney failure and a decreased chance of survival after hematopoietic-cell transplantation. There are no effective antiviral treatments for this disease.

Despite being the second most common cause of clinical disease hematopoietic-cell transplantation, very little is known about this virus. To address this knowledge gap, the investigators aim to study patients with confirmed BK virus disease post allogeneic hematopoietic-cell transplantation.

As part of this study, regular urine and blood tests will be done to understand how the virus behaves over time and which organs it affects. Blood and urine samples will also be obtained to study how the immune system rebuilds itself after hematopoietic-cell transplantation. Finally, an ultrasound of the kidneys and the bladder will be done to evaluate for any presence of disease in these organs.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥18 years old
* All adult patients who undergo allo-HCT will be eligible for the study, regardless of age, underlying disease, conditioning regimen, or GVHD prophylaxis regimen

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients who undergo allo-HCT will be eligible for the study, regardless of age, underlying disease, conditioning regimen, or GVHD prophylaxis regimen
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
The mean total number of cytokine producing BKV-specific NK and T-cells at the time of BKVD in affected patients, as compared with unaffected patients | 2 years

SECONDARY OUTCOMES:
Analytically determine a BKV-specific cfDNA methylation pattern in the urine and plasma samples of affected patients | 2 years
Analytically determine BKV-specific antibody glycosylation patterns in plasma samples of patients who exhibit BKVR. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Ritz, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No